CLINICAL TRIAL: NCT02471482
Title: Effect of Mozart Music on Cerebral Oxygenation and Behavioural Response of Premature Infants Between 28-32 Weeks of Corrected Gestation
Brief Title: Effect of Mozart Music on Cerebral Oxygenation and Behavioural Response of Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Principal Investigator, Faiza Yasin, Dr, Coombe Women and Infants University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Study No. 6 - 2013
Record Dates: First submitted 2014-11-07; First posted 2015-06-15 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Premature Brain Oxygenation
Keywords: Near Infra Red Spectrometry; Cerebral oxygenation; Mozart music
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music First group (Experimental): Mozart music lullaby for 30 minutes with recording of cerebral oxygenation (by using Near infrared spectroscopy) and vital signs (respiratory rate, heart rate, oxygen saturations and frequency of apneic episodes continuously) followed by 10 minutes of "washout" period and then period of no music for next 30 minutes (with same variables recorded as outlined for music session).
  This cycle is repeated every 6 hours for 24 hours. In addition, the behavioral response of baby is observed during the study period by video recording which will be in 'Mute' video mode and then reviewed by our developmental staff
  Interventions: Other: Mozart music lullaby
- No Music First group (Experimental): No music in first 30 minutes of study followed by 10 minutes of "washout" period and then 30 minutes of Mozart music lullaby while recording same variables. This cycle was repeated every 6 hours for 24 hours.
  Interventions: Other: Mozart music lullaby

INTERVENTIONS:
Other: Mozart music lullaby — Recorded Mozart Lullaby will be played. The noise level will be kept below 45db as recommended by American Academy of Pediatrics and will be monitored by sound monitor placed in incubator during the study period. Enrolled babies will have hearing screening performed prior to discharge from hospital.
  Other Names: Music

SUMMARY:
This study is intended to see the effect of Mozart music on oxygen content of brain of premature infants once they achieve corrected gestation of 28-32 weeks and are clinically stable. Each baby is its own control. Difference of Oxygenation of brain will be measured during period with and without music. In addition behavioural response of baby will be recorded during intervention

DETAILED DESCRIPTION:
Study Group:

Stable Infants of corrected age of 28-32weeks will be enrolled at more than seven days age according to inclusion criteria.

An informed written consent will be obtained from parents/guardians after providing information leaflet and verbal explanation.

INCLUSION CRITERIA:

* Babies with corrected age of 28-32(28+0 to32+0) weeks of gestation, more than seven days old
* Breathing spontaneously in room air or stable on nCPAP with FiO2 requirement less than 30%
* Not requiring inotropic support
* On full enteral feeds.

EXCLUSION CRITERIA:

* Babies with major congenital abnormalities
* Intraventricular haemorrhage grade 3 and 4 or cystic periventricular leucomalacia on cranial ultrasound

Study Design:

A randomized crossover study will be conducted in tertiary care level at Coombe Women and Infants University Hospital, Dublin.

As this is a randomized crossover study, each baby will act as his/her own control. Enrolled babies will be randomized to 'Music' or 'No Music'. All babies will be studied one hour after feed. The baby randomized to 'Music' will be played music for 30 minutes with recording of cerebral oxygenation (by using Near infrared spectroscopy) and vital signs (respiratory rate, heart rate, oxygen saturations and frequency of apneic episodes every 10 minutes) followed by 10 minutes of "washout" period and then period of no music for next 30 minutes (with same variables recorded as outlined for music session).

Baby randomized to 'No Music' will have no music in first 30 minutes of study followed by 10 minutes of "washout" period and then 30 minutes of music. This cycle will be repeated every 6 hours for 24 hours.

In addition the investigators will observe the behavioral response of baby during the study period by video recording which will be 'Mute' video recorded and then reviewed by our developmental staff. The behavior will be documented on 'Neonatal Behavioral Observation Sheet'. The observations will include, in addition to vital signs, the facial expression, posture and motor responses of baby during phases of music and no music.

The investigators plan to blind the study to the medical staff and also to the researchers at the time of the study (using research blind mode on near infrared spectroscopy machine). In this mode the data are stored, however not displayed at the time of the study.

Recorded Mozart Lullaby will be played. The noise level will be kept below 45db as recommended by American Academy of Pediatrics and will be monitored by sound monitor placed in incubator during the study period. Enrolled babies will have hearing screening performed prior to discharge from hospital.

Randomization: Sealed opaque envelopes

Music:

The music used will be Mozart Lullaby. This will be played on a small MP3 that will be placed baby's incubator 5cm away from baby's head. The noise level is aimed to be kept under 45dB as per hospital recommendation by adjusting volume of MP3 player. TheMP3 player will be covered in a clean plastic bag for hygiene purpose. The background will be kept to minimum during the study period.

Statistical analysis:

Statistical analysis will be performed using the SPSS software, V.17. Data will be analyzed by t-test to determine significant difference of cerebral blood flow during phase with and without music. Significance will be defined as p<0.05. As there are no data for normal brain oxygenation for the cohort studied, the investigators plan to enroll 30 infants in the pilot phase.

ELIGIBILITY:
Inclusion Criteria:

* Babies with corrected age of 28-32(28+0 to32+0) weeks of gestation, more than seven days old
* Breathing spontaneously in room air or stable on nCPAP with FiO2 requirement less than 30%
* Not requiring inotropic support
* On full enteral feeds.

Exclusion Criteria:

* Babies with major congenital abnormalities
* Intraventricular haemorrhage grade 3 and 4 or cystic periventricular leucomalacia on cranial ultrasound

Ages: 7 Days to 35 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in cerebral oxygenation values with and without Mozart music as assessed by near infra red spectroscopy | One hour after feeding, period of music (assessed up to 30 minutes), wash out period (assessed in next 10 minutes), period of no music (assessed in next 30 minutes). Same cycle would be repeated every six hours for 24 hours only.
  Using Near infra red spectroscopy electrodes placed over baby's scalp

SECONDARY OUTCOMES:
Heart rate | One hour after feeding, period of music (assessed up to 30 minutes), wash out period (assessed in next 10 minutes), period of no music (assessed in next 30 minutes). Same cycle would be repeated every six hours for 24 hours only.
  Recorded every minute using continuous stream monitoring by bed master
Respiratory rate | One hour after feeding, period of music (assessed up to 30 minutes), wash out period (assessed in next 10 minutes), period of no music (assessed in next 30 minutes). Same cycle would be repeated every six hours for 24 hours only.
  Recorded every minute using continuous stream monitoring by bed master
Oxygen saturation | One hour after feeding, period of music (assessed up to 30 minutes), wash out period (assessed in next 10 minutes), period of no music (assessed in next 30 minutes). Same cycle would be repeated every six hours for 24 hours only.
  Recorded every minute using continuous stream monitoring by bed master
Apnea episode | One hour after feeding, period of music (assessed up to 30 minutes), wash out period (assessed in next 10 minutes), period of no music (assessed in next 30 minutes). Same cycle would be repeated every six hours for 24 hours only.
  Recorded every minute using continuous stream monitoring by bed master
Behavioural response to Mozart music | One hour after feeding, period of music (assessed up to 30 minutes), wash out period (assessed in next 10 minutes), period of no music (assessed in next 30 minutes). Same cycle would be repeated every six hours for 24 hours only.
  Continuous video made and later assessed by two developmental nurses and using Newborn Individualized Developmental Care and Assessment Program (NIDCAP)/observation sheet. Both nurses were blinded for time of music as video was mute.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Yasin, Principal Investigator — Neonatal Department, Coombe Women and Infants University Hospital, Dublin-8,Ireland